CLINICAL TRIAL: NCT03242577
Title: An Exploratory Comparative Pilot Study to Identify the Most Appropriate Method for Microbial Consortia Sampling From the Skin-II
Brief Title: Micro-Technique Sampling
Status: Completed | Type: Observational
Sponsor: Kimberly-Clark Corporation (Industry)
Responsible Party: Sponsor
Other Study IDs: 500-17-07
Record Dates: First submitted 2017-08-03; First posted 2017-08-08 (Actual); Last update posted 2017-11-01 (Actual); Status verified 2017-10

CONDITIONS: Dermatitis
MeSH Terms: conditions — Dermatitis

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This is a single-center, exploratory comparative pilot study to identify the most appropriate method for microbial consortia sampling from the skin.

Ten subjects are expected to complete the study at one investigative site in the United States.

The study will consist of 2 visits, Visit 1 (Screening), Visit 2 (Sampling). At Visit 1, subjects will be consented and have their eligibility reviewed. Visit 1 and Visit 2 may be combined into one visit. Visit 1 will involve the informed consent process, screening, and enrollment. Visit 2 will involve sampling of eight (8) test sites on the back with three (3) different sampling methods: swabbing (2 sites/method), cup scrub (2 sites/method), and tape stripping (4 sites/method). All samples will be returned to Kimberly Clark then sent to a laboratory for analysis.

ELIGIBILITY:
Inclusion Criteria:

* Fluent in English, willing and able to read, understand, and sign the informed consent form (ICF);
* Ability to complete the course of the study and comply with instructions;
* Females aged 18 to 40 years, in good general health as deemed by the investigator (no physical required);
* Individuals free of any systemic or dermatological disorder, tatoos in the testing area or recent tanning bed exposure
* Anticipated ability to complete the course of the study and to comply with instructions;
* Females practicing an acceptable method of birth control
* Caucasian individuals with Fitzpatrick skin type I, II, or III

Ages: 18 Years to 40 Years | Sex: Female
Age Groups: Adult
Study Population: Subjects will consist of ten (10)Caucasian female adults 18-40 years of age, at 1 US site.
Sampling Method: Probability Sample
Enrollment: 10 (Actual)
Dates: Start 2017-08-01 (Actual); Primary Completion 2017-08-02 (Actual); Study Completion 2017-08-02 (Actual)

PRIMARY OUTCOMES:
Best method for collecting skin microbiome samples | 1 day
  Composition of skin microbiome by 16SrRNA pyrosequencing from 3 skin collection methods: Swabbing; Cup Scrub; and Tape Stripping

CONTACTS AND LOCATIONS:
Overall Officials: Barry Reece, Principal Investigator — RCTs
Locations (1):
- Reliance Clinical Testing Services, Irving, Texas, United States

IPD SHARING:
Plan to Share IPD: No
Subjects will be identified on logs and other documents submitted to the Sponsor by their unique identification number with or without their initials, not by name. Documents that identify the subject (e.g., the signed informed consent) are not to be submitted to the Sponsor and must be maintained in confidence by the Investigator.